CLINICAL TRIAL: NCT02127177
Title: Long-term Effects of Continuous Positive Airway Pressure on Lipidemia and High-sensitivity C-reactive Protein Levels in Nonobese Patients With Coronary Heart Disease and Obstructive Sleep Apnea
Brief Title: Long-term Effects of CPAP on Lipidemia and Hs-CRP Levels in OSA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF2009
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Obstructive Sleep Apnea; Coronary Heart Disease
Keywords: obstructive sleep apnea; coronary heart disease; continuous positive airway pressure; lipid profiles; high-sensitivity C-reactive protein
MeSH Terms: conditions — Sleep Apnea, Obstructive; Coronary Disease | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cpap (Experimental)
  Interventions: Device: Continuous Positive Airway Pressure Ventilator
- No Cpap (No Intervention)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure Ventilator — CPAP group received fixed-level CPAP titration using an automated pressure setting device for one night. The optimal CPAP pressure for each patient in the CPAP group was set at the minimum pressure required to abolish snoring, obstructive respiratory events, and airflow limitation for 95% of the night, according to a previous validation by our study.
  Other Names: Continuous Positive Airway Pressure(CPAP)
  Arms: Cpap

SUMMARY:
The increased risk of atherosclerotic morbidity and mortality in patients with obstructive sleep apnea (OSA) has been linked to hypertension, insulin resistance, dyslipidemia, and systemic inflammation. The relationship regarding obstructive sleep apnea (OSA) and lipidemia and systemic inflammation is far from conclusion for obesity as a strong confounding factor.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep disorder characterized by recurrent episodes of partial or complete obstruction of the upper airway during sleep, resulting in sleep fragmentation and oxyhemoglobin desaturation. OSA is recognized as an important public health problem in developed country, affecting 9 and 24% of middle-aged females and males, respectively. OSA, however, is not recognized as an abnormality for the majority and doesn't get more attention from most people in China. Increasing evidence now indicates that severe OSA is associated with increased cardiovascular morbidity and mortality, mainly due to acute myocardial infarction and stroke. Atherosclerosis is a key mechanism for these cardiovascular events. Numerous studies have explored the relationship between hypertension and OSA. And these studies confirms that OSA is an important identifiable cause of hypertension and a raised blood pressure has been shown to fall with effective continuous positive airway pressure (CPAP) treatment. Dyslipidemia, an established independent risk factor for coronary heart disease (CHD) and atherosclerosis, is common in patients with OSA. But there are limited interventional data on OSA and lipidemia, showing controversial results. Several studies9,10 have shown a direct relationship between OSA and lipid profiles, independently of obesity, while other studies have demonstrated that obesity, as a confounding factor, contributed to dyslipidemia among OSA patients.11,12 Taken together, adiposity is a strong confounding factor for interpretation of the causal relationship between dyslipidemia and OSA. Few studies have focused on nonobese patients.10,13 There are only a small number of randomized trials that have examined the effect of CPAP on fasting lipid profiles14,15 and none were specifically designed to evaluate the lipid profiles. Furthermore, most studies assessed the impact of CPAP on OSA-related lipids without statin therapy. In this way, it may be useful to avoid the disturb conditions due to statin treatment. But it is impractical to those patients with OSA and CHD. Since statins, in addition to decreasing hyperlipidemia levels, also inhibit inflammatory cytokines and play a critical role of plaque stabilization in CHD patients. Similarly, the condition existed in the examination of high-sensitivity C-reactive protein (hs-CRP) in CHD subjects with OSA. Therefore, the aims of the present study were (1) to establish whether CPAP therapy decreases lipid profiles and hs-CRP levels in nonobese patients with CHD and OSA, (2) to establish whether a relationship exists between the severity of OSA and levels of these circulating markers, and (3) to demonstrate a possible mechanism for the prevention of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with a confirmation of CHD and moderate to severe

Exclusion Criteria:

* A body mass index (BMI) ≥ 25 kg/m2
* Established hypertension, diabetes mellitus, predominantly central sleep apnea, hypothyroidism
* A history of smoking, chronic obstructive pulmonary disease, atopy, rhinitis, arthritis
* Pharmacological treatment that could affect lipids and hs-CRP levels
* Epworth Sleepiness Scale (ESS) ≥15
* Diagnosed with malignant cancer with a life expectancy of less than 1 years
* Severe psychiatric disease, sustained excessive alcohol use, New York Heart Association Class III-IV degree
* Declined to participate or were unable to give informed consent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
lipid profiles | baseline, Change from baseline lipids at 6 months，Change from baseline lipids at 12 months
  plasma fasting lipid profiles were measured at baseline, 6months，and 12months.

SECONDARY OUTCOMES:
High-sensitivity C-reactive protein | baseline,Change from baseline high-sensitivity C-reactive protein at 6 months,Change from baseline high-sensitivity C-reactive protein at 12 months
  Fasting plasma high-sensitivity C-reactive protein was analyzed at baseline,6 months,and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- center of pulmonary vascular disease, Fuwai hospital, Beijing, China

REFERENCES:
- [Derived] Huang Z, Liu Z, Zhao Z, Zhao Q, Luo Q, Tang Y. Effects of Continuous Positive Airway Pressure on Lipidaemia and High-sensitivity C-reactive Protein Levels in Non-obese Patients with Coronary Artery Disease and Obstructive Sleep Apnoea. Heart Lung Circ. 2016 Jun;25(6):576-83. doi: 10.1016/j.hlc.2015.10.021. Epub 2016 Jan 4. PMID 26804247